CLINICAL TRIAL: NCT01842243
Title: Multiparametric CMR Assessment of Apical Versus Septal Pacing Study
Brief Title: Effect of Septal Versus Apical Pacing- a Comparative Study Using Cardiac MRI
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Abbott Medical Devices (Industry); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2011CD016
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2013-01

CONDITIONS: Ventricular Dysfunction; Ventricular Remodelling
Keywords: Ventricular dysfunction; MRI; Echocardiography; Pacemakers
MeSH Terms: conditions — Ventricular Dysfunction; Ventricular Remodeling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apical Pacing (Active Comparator): Pacemaker programmed to pacing the heart at apex for 9 months.
  Interventions: Procedure: Apical pacing; Procedure: Septal pacing; Device: Pacemaker
- Septal Pacing (Active Comparator): Pacemaker programmed to pacing the heart at the septum for 9 months.
  Interventions: Procedure: Apical pacing; Procedure: Septal pacing; Device: Pacemaker

INTERVENTIONS:
Procedure: Apical pacing — Pacemaker set to pace at right ventricular apex initially.
Procedure: Septal pacing — Pacemaker set to pace at right ventricular septum initially.
Device: Pacemaker — MR conditional Pacemaker implanted in all study patients
  Other Names: MR conditional Pacemaker

SUMMARY:
Despite considerable effort the optimal site to place a pacemaker lead at the time of pacemaker implant remains unclear. Historically pacemaker leads have always been inserted at the bottom (apex) of the heart. It is suggested that a lead placed at the apex is associated with an increase in heart rhythm problems and also heart failure (impaired pumping function). The top of the ventricle (septum) has been investigated as an alternative site and is now routinely used by some centres. Previous estimation of the hearts pumping function (ejection fraction) has been limited to the use of echo (sound waves). Echo is not sensitive enough to detect small changes in the ejection fraction reliably (measure of pumping function of heart). The gold standard for measurement of ejection fraction is MRI (using magnets). Previous pacemakers have not been compatible with MRI scans. The latest generation of pacemakers are now able to be safely scanned within an MRI scanner. This allows a much more accurate estimation of the effects of a pacemaker on the ejection fraction which has not yet been studied.

The investigators plan to study those patients undergoing a pacemaker implant and ablation procedure as part of their standard care.

Individuals will have an exercise test, blood test used to measure biomarkers and fill in a symptom questionnaire.

Individuals will have a Cardiac MR compatible pacemaker fitted and 2 ventricular leads will be inserted, one apically and one septally. Only one lead will be used at any given time. Individuals will then undergo their planned AV node ablation.

Following this they will have a cardiac MR scan. Further MRI scans will be performed at 9 and 18 month intervals, as will symptom questionnaires, blood tests (BNP) to determine heart muscle strain, exercise testing and echocardiograms.

The hypothesis is that a lead placed on the septum will produce superior cardiac performance over the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients in permanent Atrial Fibrillation (AF)requiring a pacemaker on clinical grounds (tachycardia/bradycardia syndrome or requiring an AV node ablation)and AV node ablation or a pacemaker for rate control)
* Patients aged 18 to 85 years old.
* Able to consent for study.

Exclusion Criteria:

* Patients with moderate to severe LV dysfunction (EF < 40%).
* Any contraindication to an MRI scan.
* Patients indicated for an Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy.
* Patients with a Myocardial Infarction within three months prior to enrollment.
* Patients that received bypass surgery within three months prior to enrollment.
* Patients that had a valve replacement within three months prior to enrollment or patients with a mechanical right heart valve.
* Patients where a right ventricular lead cannot be placed e.g. complex congenital heart disease.
* Patients with hypertrophic obstructive cardiomyopathy.
* Patients with acute coronary syndrome, unstable angina, severe mitral regurgitation and/or haemodynamically significant aortic stenosis.
* Previous implanted pacemaker or cardioverter defibrillator.
* Terminal conditions with a life expectancy of less than two years.
* Participation in any other study that would confound the results of this study.
* Psychological or emotional problems that may interfere with the volunteer's ability to provide full consent or fully understand the purposes of the study.
* Pregnant patients or patients who may become pregnant during the time-scale of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Ventricular Ejection fraction | 18 months
  Comparison of % change in Left and Right Ventricular Ejection Fractions between apical and septal pacing groups as measured on MRI.

SECONDARY OUTCOMES:
Levels of BNP | 18 months
  Blood Sampling
MRI measures of Left and Right ventricular dyssynchrony | 18 months
Exercise Capacity as measured by CPEX | 18 months
6 minute walk tests | 18 months
Quality of life measures SF36 | 18 months
Level of Pro-BNP | 18 months
  Blood sampling
Level of ICTP | 18 months
  Blood sampling
Level of MMP-1 | 18 months
  Blood sampling
Level of MMP2 | 18 months
  Blood sampling
Level of MMP-9 | 18 months
  Blood sampling
Level of Troponin | 18 months
  Blood sampling
Level of GDF-15 | 18 months
  Blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dr Ainslie, MBChB, Principal Investigator — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester NHS trust, Manchester, United Kingdom